CLINICAL TRIAL: NCT01175083
Title: Immunogenicity, Safety and Reactogenicity of GSK Biologicals' Pneumococcal Vaccine 1024850A When Administered to Children Between 8 Weeks and 2 Years of Age
Brief Title: Immunization of Children Between 8 Weeks and 2 Years of Age With GSK Pneumococcal Vaccine GSK1024850A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114056; 2012-000254-64 (EudraCT Number)
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-02

CONDITIONS: Infections, Streptococcal
Keywords: Immunogenicity; Booster vaccination; Catch-up vaccination; Pneumococcal vaccine; Pneumococcal disease; Sickle cell disease; Safety
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections; Anemia, Sickle Cell | interventions — PHiD-CV vaccine

ARMS (6):
- Tritanrix-HepB/Hib+Polio Sabin <6S Group (Experimental): Children below (<) 6 months of age at time of enrolment, diagnosed with sickle cell disease (S), who received a 3-dose primary vaccination at Study Months 0, 1 and 2 with Synflorix vaccine co-administered with Tritanrix-HepB/Hib and Polio Sabin vaccines, followed by a booster vaccination at Study Month 8.
  Interventions: Biological: GSK1024850A (Synflorix); Biological: Tritanrix-HepB/Hib; Biological: Polio Sabin
- Tritanrix-HepB/Hib+Polio Sabin <6NS Group (Active Comparator): Healthy children, below (<) 6 months of age at time of enrolment, who received a 3-dose primary vaccination at Study Months 0, 1 and 2 with Synflorix vaccine co-administered with Tritanrix-HepB/Hib and Polio Sabin vaccines, followed by a booster vaccination at Study Month 8.
  Interventions: Biological: GSK1024850A (Synflorix); Biological: Tritanrix-HepB/Hib; Biological: Polio Sabin
- Synflorix 7-11S Group (Experimental): Children between 7-11 months of age at time of enrolment, diagnosed with sickle cell disease (S), who received a 2-dose primary vaccination at Study Months 0 and 1 with Synflorix vaccine, followed by a booster vaccination at Study Month 3.
  Interventions: Biological: GSK1024850A (Synflorix)
- Synflorix 7-11NS Group (Active Comparator): Healthy children between 7-11 months of age at time of enrolment, who received a 2-dose primary vaccination at Study Months 0 and 1 with Synflorix vaccine, followed by a booster vaccination at Study Month 3.
  Interventions: Biological: GSK1024850A (Synflorix)
- Synflorix 12-23S Group (Experimental): Children between 12-23 months of age at time of enrolment, diagnosed with sickle cell disease (S), who received a 2-dose vaccination with Synflorix vaccine, at Study Months 0 and 2.
  Interventions: Biological: GSK1024850A (Synflorix)
- Synflorix 12-23NS Group (Active Comparator): Healthy children between 12-23 months of age at time of enrolment, who received a 2-dose vaccination with Synflorix vaccine, at Study Months 0 and 2.
  Interventions: Biological: GSK1024850A (Synflorix)

INTERVENTIONS:
Biological: GSK1024850A (Synflorix) — 2, 3 or 4 intramuscular injection
Biological: Tritanrix-HepB/Hib — Intramuscular injection, 4 doses
  Other Names: DTPw-HBV/Hib
  Arms: Tritanrix-HepB/Hib+Polio Sabin <6NS Group; Tritanrix-HepB/Hib+Polio Sabin <6S Group
Biological: Polio Sabin — 4 oral doses
  Other Names: OPV
  Arms: Tritanrix-HepB/Hib+Polio Sabin <6NS Group; Tritanrix-HepB/Hib+Polio Sabin <6S Group

SUMMARY:
The aim of the study is to evaluate the immunogenicity, safety and reactogenicity of GSK Biologicals' pneumococcal conjugate vaccine GSK1024850A.

Children that are below 6 months at the time of enrolment will also receive the DTPw-HBV/Hib and OPV vaccines.

DETAILED DESCRIPTION:
This protocol posting has been updated according to Protocol Amendment 2, September 2010. The impacted sections are arms and inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* A male or female between, and including:

  * 8 and 11 weeks of age at the time of the first vaccination for subjects in the <6S and <6NS groups or
  * 7 and 11 months at the time of the first vaccination for subjects in the 7-11S and 7-11NS groups or
  * 12 and 23 months at the time of first vaccination for subjects in the 12-23S and 12-23NS groups (Note the second dose should be administered at 23 Months of age at the latest to allow, if needed, compliance with the National Recommendations on administration of the 23-valent polysaccharide pneumococcal vaccine in children with SCD as of 24 months of age).
* Written informed consent, signed or thumb printed, obtained from the parent(s)/LAR(s) of the subject. Where parent(s)/LAR(s) are illiterate, the consent form will be countersigned by a witness.

Additional inclusion criteria for children with SCD (<6S, 7-11S and 12-23S groups):

* Children with diagnosis of sickle cell disease [homozygous sickle cell disease (hemoglobin SS disease), double heterozygous sickle hemoglobin C disease (hemoglobin SC disease) and the sickle ß-thalassemias] and confirmed hemoglobin status by hemoglobin chromatography and electrophoresis (<6S group) or electrophoresis (7-11S and 12-23S groups).
* Free of any other known or suspected health problems (as established by medical history and clinical examination before entering into the study), that would contraindicate the initiation of routine immunizations outside a clinical trial context

Additional inclusion criteria for healthy children (<6NS, 7-11NS and 12-23NS groups):

* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Children with negative diagnosis of sickle cell disease and confirmed hemoglobin status by hemoglobin chromatography and/or electrophoresis.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of study vaccines and ending 30 days after. Locally recommended vaccines (recommended through the EPI program or through national immunization campaigns) for example inactivated influenza vaccine are always allowed, even if concomitantly administered with the study vaccines, but should be documented in the eCRF.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous vaccination or planned vaccination during the study with any pneumococcal vacccine.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital malformations.
* History of any neurological disorders or seizures.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Birth weight below 1500g.
* Serious chronic illness other than SCD.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C on oral, axillary or tympanic setting, or ≥ 38.0°C on rectal setting. The preferred route for recording temperature in this study will be tympanic.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.

Additional exclusion criteria for children with SCD (<6S, 7-11S and 12-23S groups):

• Any confirmed or suspected immunosuppressive or immunodeficient condition, (including human immunodeficiency virus (HIV) infection) other than SCD related conditions, based on medical history and physical examination (no laboratory testing required).

Additional exclusion criteria for healthy children (<6 NS, 7-11NS and 12-23NS groups):

• Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, based on medical history and physical examination (no laboratory testing required).

Ages: 8 Weeks to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2013-01-17 (Actual); Study Completion 2013-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Sirima SB, Tiono A, Gansane Z, Siribie M, Zongo A, Ouedraogo A, Francois N, Strezova A, Dobbelaere K, Borys D. Immunogenicity and Safety of 10-valent Pneumococcal Nontypeable Haemophilus influenzae Protein D Conjugate Vaccine (PHiD-CV) Administered to Children With Sickle Cell Disease Between 8 Weeks and 2 Years of Age: A Phase III, Open, Controlled Study. Pediatr Infect Dis J. 2017 May;36(5):e136-e150. doi: 10.1097/INF.0000000000001518. PMID 28403055
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Primary Epoch
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Started | 50 | 50 | 50 | 50 | 50 | 50
Completed | 50 | 50 | 50 | 50 | 50 | 47
Not Completed | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Period: Booster Epoch
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Started | 49 (One subject died between both Epochs and hence did not participate in the Booster Epoch.) | 49 (One subject died between both Epochs and hence did not participate in the Booster Epoch.) | 50 | 50 | 0 (No subjects participated in the Booster Epoch, as no booster dose was planned per protocol.) | 0 (No subjects participated in the Booster Epoch, as no booster dose was planned per protocol.)
Completed | 49 | 49 | 49 | 49 | 0 | 0
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group | Total
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50 | 300
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.4 (0.9) | 8.6 (0.9) | 8.6 (1.5) | 8.3 (1.2) | 16.6 (3.3) | 16.7 (3.5) | 11.2 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 29 | 26 | 32 | 15 | 24 | 147
  Male | 29 | 21 | 24 | 18 | 35 | 26 | 153
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage/African American | 50 | 50 | 50 | 50 | 50 | 50 | 300

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes for Subjects Receiving Synflorix Vaccine Co-administered With Tritanrix-HepB/Hib and Polio Sabin Vaccines
Description: Antibodies have been assessed against the following vaccine pneumococcal serotypes: 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (µg/mL). The seropositivity cut-off of the assay was an antibody concentration greater than or equal to (≥) 0.05 micrograms per milliliter (µg/mL). Antibody concentrations below than (<) 0.05 µg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: One month after primary vaccination (Month 3)
Population: The analysis was performed on the According To Protocol (ATP) immunogenicity cohort and included all subjects who were co-administered Synflorix with Tritanrix-HepB/Hib and Polio Sabin vaccines, for whom data concerning immunogenicity outcomes and assay results for antibodies against at least one vaccine antigen component were available at Month 3.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 48 | 46
µg/mL
  Anti-1 | 3.51 [2.77 to 4.44] | 3.63 [2.91 to 4.53]
  Anti-4: number analyzed (Participants) | 47 | 46
  Anti-4 | 4.25 [3.18 to 5.67] | 3.51 [2.73 to 4.51]
  Anti-5: number analyzed (Participants) | 47 | 46
  Anti-5 | 5.15 [4.07 to 6.51] | 5.94 [4.91 to 7.18]
  Anti-6B | 1.29 [0.83 to 1.99] | 1.13 [0.74 to 1.72]
  Anti-7F | 4.91 [3.84 to 6.28] | 4.28 [3.49 to 5.26]
  Anti-9V: number analyzed (Participants) | 47 | 46
  Anti-9V | 4.56 [3.51 to 5.92] | 4.59 [3.70 to 5.70]
  Anti-14: number analyzed (Participants) | 46 | 46
  Anti-14 | 4.30 [3.08 to 6.00] | 5.95 [4.27 to 8.29]
  Anti-18C: number analyzed (Participants) | 47 | 45
  Anti-18C | 14.60 [11.01 to 19.36] | 11.33 [8.47 to 15.17]
  Anti-19F: number analyzed (Participants) | 47 | 46
  Anti-19F | 11.87 [9.05 to 15.57] | 9.78 [7.01 to 13.64]
  Anti-23F | 1.32 [0.90 to 1.93] | 1.41 [0.95 to 2.11]

2. Primary Outcome: Concentrations of Antibodies Against Protein D (PD) for Subjects Receiving Synflorix Vaccine Co-administered With Tritanrix-HepB/Hib and Polio Sabin Vaccines
Description: Anti-PD antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 100 EL.U/mL. Antibody concentrations < 100 EL.U/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: One month after the primary vaccination (Month 3)
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who were co-administered Synflorix with Tritanrix-HepB/Hib and Polio Sabin vaccines, for whom data concerning immunogenicity outcomes and assay results for antibodies against at least one vaccine antigen component were available at Month 3.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 47 | 46
EL.U/mL | 2789.09 [2313.89 to 3361.87] | 3065.40 [2530.54 to 3713.31]

3. Secondary Outcome: Concentration of Antibodies Against Vaccine Pneumococcal Serotypes for Subjects Receiving Synflorix Vaccine Co-administered With Tritanrix-HepB/Hib and Polio Sabin Vaccines
Description: Antibodies have been assessed against the following vaccine pneumococcal serotypes: 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (µg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 micrograms per milliliter (µg/mL). Antibody concentrations < 0.05 µg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: Prior to the primary vaccination (Month 0), prior to (Month 8) and one month after (Month 9) booster vaccination
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who were co-administered Synflorix with Tritanrix-HepB/Hib and Polio Sabin vaccines, for whom data concerning immunogenicity outcomes and assay results for antibodies against at least one vaccine antigen component were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 48 | 46
μg/mL
  Anti-1, Month 0: number analyzed (Participants) | 46 | 42
  Anti-1, Month 0 | 0.09 [0.06 to 0.12] | 0.09 [0.06 to 0.12]
  Anti-1, Month 8: number analyzed (Participants) | 44 | 38
  Anti-1, Month 8 | 0.67 [0.54 to 0.84] | 0.69 [0.52 to 0.90]
  Anti-1, Month 9: number analyzed (Participants) | 44 | 38
  Anti-1, Month 9 | 5.34 [4.07 to 7.02] | 5.14 [3.52 to 7.50]
  Anti-4, Month 0: number analyzed (Participants) | 48 | 45
  Anti-4, Month 0 | 0.04 [0.03 to 0.06] | 0.06 [0.04 to 0.08]
  Anti-4, Month 8: number analyzed (Participants) | 44 | 38
  Anti-4, Month 8 | 1.20 [0.91 to 1.59] | 1.08 [0.77 to 1.52]
  Anti-4, Month 9: number analyzed (Participants) | 44 | 38
  Anti-4, Month 9 | 7.04 [5.53 to 8.97] | 6.02 [4.40 to 8.24]
  Anti-5, Month 0 | 0.06 [0.05 to 0.09] | 0.07 [0.06 to 0.10]
  Anti-5, Month 8: number analyzed (Participants) | 44 | 38
  Anti-5, Month 8 | 1.13 [0.87 to 1.47] | 1.23 [0.93 to 1.63]
  Anti-5, Month 9: number analyzed (Participants) | 43 | 37
  Anti-5, Month 9 | 6.30 [4.94 to 8.04] | 6.91 [4.92 to 9.73]
  Anti-6B, Month 0: number analyzed (Participants) | 47 | 40
  Anti-6B, Month 0 | 0.07 [0.05 to 0.09] | 0.11 [0.07 to 0.18]
  Anti-6B, Month 8: number analyzed (Participants) | 44 | 38
  Anti-6B, Month 8 | 1.94 [1.55 to 2.44] | 1.62 [1.25 to 2.09]
  Anti-6B, Month 9: number analyzed (Participants) | 44 | 37
  Anti-6B, Month 9 | 5.07 [4.16 to 6.18] | 5.00 [3.71 to 6.74]
  Anti-7F, Month 0: number analyzed (Participants) | 47 | 44
  Anti-7F, Month 0 | 0.08 [0.06 to 0.11] | 0.13 [0.09 to 0.19]
  Anti-7F, Month 8: number analyzed (Participants) | 44 | 38
  Anti-7F, Month 8 | 1.83 [1.41 to 2.37] | 1.57 [1.21 to 2.05]
  Anti-7F, Month 9: number analyzed (Participants) | 44 | 38
  Anti-7F, Month 9 | 9.03 [7.18 to 11.37] | 8.19 [6.18 to 10.86]
  Anti-9V, Month 0: number analyzed (Participants) | 47 | 44
  Anti-9V, Month 0 | 0.12 [0.08 to 0.16] | 0.12 [0.09 to 0.16]
  Anti-9V, Month 8: number analyzed (Participants) | 44 | 38
  Anti-9V, Month 8 | 1.61 [1.17 to 2.21] | 1.44 [1.13 to 1.82]
  Anti-9V, Month 9: number analyzed (Participants) | 44 | 38
  Anti-9V, Month 9 | 8.19 [6.61 to 10.14] | 7.95 [5.94 to 10.63]
  Anti-14, Month 0: number analyzed (Participants) | 48 | 44
  Anti-14, Month 0 | 0.77 [0.53 to 1.12] | 0.65 [0.42 to 0.99]
  Anti-14, Month 8: number analyzed (Participants) | 44 | 38
  Anti-14, Month 8 | 2.58 [1.90 to 3.51] | 2.10 [1.32 to 3.34]
  Anti-14, Month 9: number analyzed (Participants) | 44 | 38
  Anti-14, Month 9 | 8.66 [6.91 to 10.85] | 7.43 [4.72 to 11.70]
  Anti-18C, Month 0: number analyzed (Participants) | 48 | 45
  Anti-18C, Month 0 | 0.13 [0.10 to 0.18] | 0.13 [0.09 to 0.18]
  Anti-18C, Month 8: number analyzed (Participants) | 44 | 38
  Anti-18C, Month 8 | 3.82 [2.97 to 4.92] | 3.16 [2.32 to 4.31]
  Anti-18C, Month 9: number analyzed (Participants) | 44 | 38
  Anti-18C, Month 9 | 16.52 [12.81 to 21.32] | 16.74 [12.98 to 21.58]
  Anti-19F, Month 0: number analyzed (Participants) | 48 | 45
  Anti-19F, Month 0 | 0.34 [0.23 to 0.51] | 0.30 [0.21 to 0.44]
  Anti-19F, Month 8: number analyzed (Participants) | 44 | 38
  Anti-19F, Month 8 | 3.31 [2.51 to 4.38] | 3.27 [2.21 to 4.84]
  Anti-19F, Month 9: number analyzed (Participants) | 44 | 38
  Anti-19F, Month 9 | 10.96 [8.37 to 14.34] | 11.27 [8.18 to 15.54]
  Anti-23F, Month 0: number analyzed (Participants) | 48 | 43
  Anti-23F, Month 0 | 0.13 [0.09 to 0.20] | 0.10 [0.07 to 0.14]
  Anti-23F, Month 8: number analyzed (Participants) | 44 | 38
  Anti-23F, Month 8 | 0.67 [0.48 to 0.94] | 0.77 [0.51 to 1.17]
  Anti-23F, Month 9: number analyzed (Participants) | 44 | 38
  Anti-23F, Month 9 | 4.86 [3.34 to 7.07] | 4.54 [2.70 to 7.62]

4. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes for Subjects Who Received a Two-dose Primary Vaccination Followed by a Booster Dose
Description: as for outcome 3
Time Frame: Prior to (Month 0) and one month after (Month 2) primary vaccination, prior to (Month 3) and one month after (Month 4) booster vaccination
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose primary vaccination followed by a booster dose, for whom data concerning immunogenicity outcomes and assay results for antibodies against at least one vaccine antigen component were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix 7-11S Group | Synflorix 7-11NS Group
Number analyzed (Participants) | 50 | 50
µg/mL
  Anti-1, Month 0: number analyzed (Participants) | 48 | 46
  Anti-1, Month 0 | 0.03 [0.03 to 0.03] | 0.04 [0.03 to 0.05]
  Anti-1, Month 2: number analyzed (Participants) | 50 | 48
  Anti-1, Month 2 | 5.48 [4.34 to 6.93] | 3.99 [3.24 to 4.91]
  Anti-1, Month 3: number analyzed (Participants) | 50 | 49
  Anti-1, Month 3 | 2.68 [2.12 to 3.39] | 2.44 [1.99 to 2.98]
  Anti-1, Month 4: number analyzed (Participants) | 49 | 48
  Anti-1, Month 4 | 5.51 [4.27 to 7.10] | 4.92 [3.74 to 6.48]
  Anti-4, Month 0: number analyzed (Participants) | 49 | 50
  Anti-4, Month 0 | 0.03 [0.03 to 0.04] | 0.03 [0.02 to 0.04]
  Anti-4, Month 2: number analyzed (Participants) | 49 | 47
  Anti-4, Month 2 | 10.88 [8.94 to 13.24] | 7.55 [6.00 to 9.50]
  Anti-4, Month 3: number analyzed (Participants) | 50 | 48
  Anti-4, Month 3 | 5.72 [4.66 to 7.03] | 4.32 [3.51 to 5.32]
  Anti-4, Month 4: number analyzed (Participants) | 49 | 48
  Anti-4, Month 4 | 9.75 [7.67 to 12.39] | 7.88 [6.28 to 9.89]
  Anti-5, Month 0: number analyzed (Participants) | 48 | 50
  Anti-5, Month 0 | 0.04 [0.03 to 0.06] | 0.06 [0.05 to 0.08]
  Anti-5, Month 2: number analyzed (Participants) | 50 | 47
  Anti-5, Month 2 | 6.76 [5.14 to 8.89] | 4.59 [3.58 to 5.88]
  Anti-5, Month 3: number analyzed (Participants) | 50 | 49
  Anti-5, Month 3 | 3.68 [2.87 to 4.73] | 3.40 [2.66 to 4.33]
  Anti-5, Month 4: number analyzed (Participants) | 49 | 48
  Anti-5, Month 4 | 7.75 [6.05 to 9.92] | 7.87 [6.02 to 10.29]
  Anti-6B, Month 0: number analyzed (Participants) | 49 | 46
  Anti-6B, Month 0 | 0.03 [0.02 to 0.03] | 0.03 [0.02 to 0.03]
  Anti-6B, Month 2: number analyzed (Participants) | 49 | 49
  Anti-6B, Month 2 | 1.61 [1.03 to 2.52] | 1.48 [1.02 to 2.13]
  Anti-6B, Month 3: number analyzed (Participants) | 50 | 49
  Anti-6B, Month 3 | 1.51 [1.06 to 2.15] | 1.35 [0.98 to 1.87]
  Anti-6B, Month 4: number analyzed (Participants) | 49 | 48
  Anti-6B, Month 4 | 3.12 [2.10 to 4.64] | 2.93 [2.17 to 3.95]
  Anti-7F, Month 0 | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.05]
  Anti-7F, Month 2: number analyzed (Participants) | 49 | 49
  Anti-7F, Month 2 | 8.51 [6.94 to 10.42] | 6.67 [5.44 to 8.19]
  Anti-7F, Month 3: number analyzed (Participants) | 50 | 49
  Anti-7F, Month 3 | 5.46 [4.37 to 6.83] | 4.68 [3.76 to 5.81]
  Anti-7F, Month 4: number analyzed (Participants) | 48 | 48
  Anti-7F, Month 4 | 11.08 [8.90 to 13.81] | 10.29 [7.92 to 13.37]
  Anti-9V, Month 0: number analyzed (Participants) | 49 | 48
  Anti-9V, Month 0 | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.05]
  Anti-9V, Month 2: number analyzed (Participants) | 49 | 49
  Anti-9V, Month 2 | 2.55 [1.86 to 3.49] | 1.67 [1.21 to 2.29]
  Anti-9V, Month 3: number analyzed (Participants) | 50 | 49
  Anti-9V, Month 3 | 1.90 [1.42 to 2.56] | 1.52 [1.16 to 2.00]
  Anti-9V, Month 4: number analyzed (Participants) | 49 | 48
  Anti-9V, Month 4 | 4.73 [3.40 to 6.58] | 3.76 [2.67 to 5.30]
  Anti-14, Month 0: number analyzed (Participants) | 47 | 48
  Anti-14, Month 0 | 0.08 [0.06 to 0.12] | 0.07 [0.05 to 0.10]
  Anti-14, Month 2: number analyzed (Participants) | 50 | 46
  Anti-14, Month 2 | 4.91 [3.48 to 6.95] | 4.81 [3.67 to 6.29]
  Anti-14, Month 3: number analyzed (Participants) | 50 | 49
  Anti-14, Month 3 | 4.71 [3.45 to 6.43] | 4.98 [4.01 to 6.20]
  Anti-14, Month 4: number analyzed (Participants) | 49 | 48
  Anti-14, Month 4 | 10.24 [7.96 to 13.18] | 10.69 [8.34 to 13.71]
  Anti-18C, Month 0: number analyzed (Participants) | 50 | 49
  Anti-18C, Month 0 | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.04]
  Anti-18C, Month 2: number analyzed (Participants) | 49 | 47
  Anti-18C, Month 2 | 12.92 [9.93 to 16.82] | 14.62 [11.61 to 18.40]
  Anti-18C, Month 3: number analyzed (Participants) | 50 | 49
  Anti-18C, Month 3 | 8.43 [6.53 to 10.88] | 11.49 [9.24 to 14.29]
  Anti-18C, Month 4: number analyzed (Participants) | 49 | 48
  Anti-18C, Month 4 | 23.57 [18.38 to 30.22] | 31.88 [25.34 to 40.11]
  Anti-19F, Month 0: number analyzed (Participants) | 49 | 48
  Anti-19F, Month 0 | 0.05 [0.04 to 0.06] | 0.04 [0.04 to 0.06]
  Anti-19F, Month 2: number analyzed (Participants) | 50 | 49
  Anti-19F, Month 2 | 11.13 [7.97 to 15.54] | 9.77 [6.16 to 15.48]
  Anti-19F, Month 3: number analyzed (Participants) | 50 | 49
  Anti-19F, Month 3 | 6.54 [4.79 to 8.92] | 7.39 [5.04 to 10.81]
  Anti-19F, Month 4: number analyzed (Participants) | 49 | 48
  Anti-19F, Month 4 | 15.59 [11.24 to 21.62] | 15.85 [10.52 to 23.89]
  Anti-23F, Month 0: number analyzed (Participants) | 48 | 48
  Anti-23F, Month 0 | 0.03 [0.03 to 0.04] | 0.04 [0.03 to 0.05]
  Anti-23F, Month 2: number analyzed (Participants) | 50 | 48
  Anti-23F, Month 2 | 1.29 [0.79 to 2.10] | 0.93 [0.60 to 1.45]
  Anti-23F, Month 3: number analyzed (Participants) | 50 | 48
  Anti-23F, Month 3 | 1.00 [0.65 to 1.56] | 1.08 [0.74 to 1.56]
  Anti-23F, Month 4: number analyzed (Participants) | 49 | 48
  Anti-23F, Month 4 | 3.11 [1.85 to 5.24] | 3.17 [2.04 to 4.91]

5. Secondary Outcome: Concentration of Antibodies Against Vaccine Pneumococcal Serotypes for Subjects Who Received a Two-dose Primary Vaccination Without Any Booster Dose
Description: as for outcome 3
Time Frame: Prior to (Month 0) the first vaccine dose, prior to (Month 2) and one month after (Month 3) the second vaccine dose
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose vaccination without any booster dose, for whom data concerning immunogenicity outcomes and assay results for antibodies against at least one vaccine antigen component were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 48 | 47
μg/mL
  Anti-1, Month 0: number analyzed (Participants) | 47 | 45
  Anti-1, Month 0 | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.05]
  Anti-1, Month 2 | 1.39 [1.07 to 1.80] | 1.49 [1.18 to 1.89]
  Anti-1, Month 3: number analyzed (Participants) | 48 | 46
  Anti-1, Month 3 | 4.67 [3.75 to 5.81] | 4.26 [3.38 to 5.37]
  Anti-4, Month 0 | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.05]
  Anti-4, Month 2: number analyzed (Participants) | 47 | 47
  Anti-4, Month 2 | 4.22 [3.23 to 5.51] | 3.74 [2.96 to 4.72]
  Anti-4, Month 3: number analyzed (Participants) | 47 | 46
  Anti-4, Month 3 | 8.87 [7.03 to 11.19] | 7.02 [5.85 to 8.43]
  Anti-5, Month 0 | 0.06 [0.05 to 0.08] | 0.08 [0.06 to 0.11]
  Anti-5, Month 2 | 1.06 [0.77 to 1.47] | 1.10 [0.83 to 1.44]
  Anti-5, Month 3: number analyzed (Participants) | 48 | 46
  Anti-5, Month 3 | 5.52 [4.23 to 7.20] | 4.07 [3.06 to 5.42]
  Anti-6B, Month 0 | 0.03 [0.03 to 0.04] | 0.04 [0.03 to 0.05]
  Anti-6B, Month 2 | 0.41 [0.28 to 0.62] | 0.34 [0.24 to 0.48]
  Anti-6B, Month 3: number analyzed (Participants) | 48 | 46
  Anti-6B, Month 3 | 1.37 [0.91 to 2.07] | 1.25 [0.87 to 1.79]
  Anti-7F, Month 0 | 0.07 [0.05 to 0.11] | 0.05 [0.04 to 0.07]
  Anti-7F, Month 2 | 2.74 [2.13 to 3.52] | 3.17 [2.56 to 3.93]
  Anti-7F, Month 3: number analyzed (Participants) | 48 | 46
  Anti-7F, Month 3 | 6.81 [5.32 to 8.70] | 6.36 [5.25 to 7.69]
  Anti-9V, Month 0 | 0.08 [0.05 to 0.12] | 0.05 [0.04 to 0.07]
  Anti-9V, Month 2 | 0.99 [0.72 to 1.34] | 0.83 [0.62 to 1.11]
  Anti-9V, Month 3: number analyzed (Participants) | 48 | 46
  Anti-9V, Month 3 | 2.35 [1.85 to 3.00] | 1.72 [1.31 to 2.25]
  Anti-14, Month 0: number analyzed (Participants) | 47 | 46
  Anti-14, Month 0 | 0.11 [0.07 to 0.16] | 0.09 [0.06 to 0.12]
  Anti-14, Month 2 | 1.87 [1.46 to 2.40] | 1.24 [0.92 to 1.66]
  Anti-14, Month 3: number analyzed (Participants) | 47 | 45
  Anti-14, Month 3 | 7.59 [5.84 to 9.87] | 5.75 [4.33 to 7.62]
  Anti-18C, Month 0 | 0.04 [0.03 to 0.06] | 0.05 [0.04 to 0.07]
  Anti-18C, Month 2 | 6.21 [4.77 to 8.10] | 6.12 [4.56 to 8.21]
  Anti-18C, Month 3: number analyzed (Participants) | 47 | 45
  Anti-18C, Month 3 | 25.52 [20.66 to 31.53] | 22.64 [18.14 to 28.26]
  Anti-19F, Month 0 | 0.06 [0.04 to 0.09] | 0.08 [0.05 to 0.12]
  Anti-19F, Month 2 | 5.88 [4.44 to 7.80] | 5.12 [3.79 to 6.94]
  Anti-19F, Month 3: number analyzed (Participants) | 48 | 46
  Anti-19F, Month 3 | 18.00 [13.97 to 23.20] | 14.46 [10.81 to 19.34]
  Anti-23F, Month 0 | 0.03 [0.03 to 0.04] | 0.05 [0.03 to 0.07]
  Anti-23F, Month 2 | 0.50 [0.32 to 0.77] | 0.35 [0.25 to 0.49]
  Anti-23F, Month 3: number analyzed (Participants) | 47 | 46
  Anti-23F, Month 3 | 1.95 [1.32 to 2.87] | 1.40 [1.05 to 1.87]

6. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes for Subjects Receiving Synflorix Vaccine Co-administered With Tritanrix-HepB/Hib and Polio Sabin Vaccines
Description: Antibody concentrations against cross-reactive pneumococcal serotypes 6A and 19A (Anti-6A, -19A) were measured by 22F enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (µg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 micrograms per milliliter (µg/mL). Antibody concentrations < 0.05 µg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: Prior to (Month 0) and one month after (Month 3) primary vaccination, prior to (Month 8) and one month after (Month 9) booster vaccination
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who were co-administered Synflorix with Tritanrix-HepB/Hib and Polio Sabin vaccines, for whom assay results for antibodies against at least one cross-reactive pneumococcal serotype were available for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 48 | 45
µg/mL
  Anti-6A, Month 0: number analyzed (Participants) | 47 | 41
  Anti-6A, Month 0 | 0.10 [0.07 to 0.14] | 0.15 [0.10 to 0.23]
  Anti-6A, Month 3: number analyzed (Participants) | 46 | 43
  Anti-6A, Month 3 | 0.12 [0.08 to 0.17] | 0.10 [0.07 to 0.13]
  Anti-6A, Month 8: number analyzed (Participants) | 37 | 30
  Anti-6A, Month 8 | 0.40 [0.27 to 0.61] | 0.18 [0.10 to 0.30]
  Anti-6A, Month 9: number analyzed (Participants) | 36 | 29
  Anti-6A, Month 9 | 0.48 [0.31 to 0.74] | 0.36 [0.23 to 0.55]
  Anti-19A, Month 0: number analyzed (Participants) | 47 | 44
  Anti-19A, Month 0 | 0.24 [0.17 to 0.36] | 0.23 [0.16 to 0.33]
  Anti-19A, Month 3 | 0.26 [0.17 to 0.39] | 0.25 [0.17 to 0.37]
  Anti-19A, Month 8: number analyzed (Participants) | 44 | 38
  Anti-19A, Month 8 | 0.23 [0.15 to 0.37] | 0.21 [0.13 to 0.35]
  Anti-19A, Month 9: number analyzed (Participants) | 44 | 37
  Anti-19A, Month 9 | 1.09 [0.65 to 1.83] | 0.85 [0.50 to 1.43]

7. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes for Subjects Who Received a Two-dose Primary Vaccination Followed by a Booster Dose
Description: as for outcome 6
Time Frame: as for outcome 4
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose primary vaccination followed by a booster dose, for whom data concerning immunogenicity outcomes and assay results for antibodies against at least one cross-reactive pneumococcal serotype were available for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 7-11S Group | Synflorix 7-11NS Group
Number analyzed (Participants) | 50 | 49
Titer
  Anti-6A, Month 0: number analyzed (Participants) | 47 | 44
  Anti-6A, Month 0 | 0.03 [0.03 to 0.04] | 0.03 [0.03 to 0.04]
  Anti-6A, Month 2: number analyzed (Participants) | 48 | 46
  Anti-6A, Month 2 | 0.18 [0.11 to 0.30] | 0.16 [0.11 to 0.24]
  Anti-6A, Month 3: number analyzed (Participants) | 50 | 47
  Anti-6A, Month 3 | 0.23 [0.14 to 0.37] | 0.22 [0.16 to 0.32]
  Anti-6A, Month 4: number analyzed (Participants) | 48 | 48
  Anti-6A, Month 4 | 0.44 [0.28 to 0.70] | 0.43 [0.30 to 0.62]
  Anti-19A, Month 0: number analyzed (Participants) | 48 | 49
  Anti-19A, Month 0 | 0.04 [0.03 to 0.06] | 0.06 [0.04 to 0.10]
  Anti-19A, Month 2 | 0.46 [0.28 to 0.76] | 0.77 [0.50 to 1.18]
  Anti-19A, Month 3: number analyzed (Participants) | 50 | 48
  Anti-19A, Month 3 | 0.44 [0.27 to 0.70] | 0.77 [0.51 to 1.17]
  Anti-19A, Month 4: number analyzed (Participants) | 49 | 49
  Anti-19A, Month 4 | 1.49 [0.93 to 2.38] | 2.35 [1.50 to 3.67]

8. Secondary Outcome: Concentration of Antibodies Against Cross-reactive Pneumococcal Serotypes for Subjects Who Received a Two-dose Primary Vaccination Without Any Booster Dose
Description: as for outcome 6
Time Frame: Prior to (Month 0) the first vaccine dose, prior to (Month 2) and one month after (Month 3) the second vaccine dose
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose vaccination without any booster dose, for whom data concerning immunogenicity outcomes and assay results for antibodies against at least one cross-reactive pneumococcal serotype were available for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 48 | 47
Titer
  Anti-6A, Month 0: number analyzed (Participants) | 45 | 44
  Anti-6A, Month 0 | 0.03 [0.03 to 0.03] | 0.04 [0.03 to 0.05]
  Anti-6A, Month 2: number analyzed (Participants) | 47 | 47
  Anti-6A, Month 2 | 0.15 [0.10 to 0.23] | 0.12 [0.08 to 0.18]
  Anti-6A, Month 3: number analyzed (Participants) | 47 | 46
  Anti-6A, Month 3 | 0.39 [0.23 to 0.66] | 0.31 [0.20 to 0.48]
  Anti-19A, Month 0: number analyzed (Participants) | 47 | 45
  Anti-19A, Month 0 | 0.06 [0.04 to 0.09] | 0.07 [0.04 to 0.11]
  Anti-19A, Month 2 | 0.77 [0.50 to 1.17] | 0.75 [0.47 to 1.19]
  Anti-19A, Month 3: number analyzed (Participants) | 48 | 46
  Anti-19A, Month 3 | 3.15 [2.13 to 4.65] | 2.79 [1.93 to 4.05]

9. Secondary Outcome: Concentration of Antibodies Against Protein D (PD) for Subjects Receiving Synflorix Vaccine Co-administered With Tritanrix-HepB/Hib and Polio Sabin Vaccines
Description: as for outcome 2
Time Frame: Prior to (Month 0) primary vaccination, prior to (Month 8) and one month after (Month 9) booster vaccination
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who were co-administered Synflorix with Tritanrix-HepB/Hib and Polio Sabin vaccines, for whom data concerning immunogenicity outcomes and assay results for antibodies against protein D were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 47 | 46
EL.U/mL
  Anti-PD, Month 0 | 64.75 [50.56 to 82.92] | 70.97 [53.71 to 93.78]
  Anti-PD, Month 8: number analyzed (Participants) | 44 | 38
  Anti-PD, Month 8 | 859.87 [681.75 to 1084.52] | 840.88 [641.50 to 1102.23]
  Anti-PD, Month 9: number analyzed (Participants) | 44 | 38
  Anti-PD, Month 9 | 2871.72 [2338.21 to 3526.96] | 3137.87 [2459.92 to 4002.68]

10. Secondary Outcome: Concentration of Antibodies Against Protein D (PD) for Subjects Who Received a Two-dose Primary Vaccination Followed by a Booster Dose
Description: as for outcome 2
Time Frame: as for outcome 4
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose primary vaccination followed by a booster dose, for whom data concerning immunogenicity outcomes and assay results for antibodies against protein D were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix 7-11S Group | Synflorix 7-11NS Group
Number analyzed (Participants) | 50 | 50
EL.U/mL
  Anti-PD, Month 0: number analyzed (Participants) | 47 | 48
  Anti-PD, Month 0 | 72.73 [57.23 to 92.42] | 88.74 [70.85 to 111.13]
  Anti-PD, Month 2 | 1313.39 [1014.30 to 1700.67] | 1489.78 [1171.98 to 1893.76]
  Anti-PD, Month 3: number analyzed (Participants) | 50 | 49
  Anti-PD, Month 3 | 932.52 [732.63 to 1186.96] | 1063.54 [844.52 to 1339.37]
  Anti-PD, Month 4: number analyzed (Participants) | 49 | 48
  Anti-PD, Month 4 | 2695.50 [2150.74 to 3378.24] | 2638.27 [2049.91 to 3395.49]

11. Secondary Outcome: Concentration of Antibodies Against Protein D (PD) for Subjects Who Received a Two-dose Primary Vaccination Without Any Booster Dose
Description: as for outcome 2
Time Frame: Prior to (Month 0) the first vaccine dose, prior to (Month 2) and one month after (Month 3) the second vaccine dose
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose vaccination without any booster dose, for whom data concerning immunogenicity outcomes and assay results for antibodies against protein D were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 48 | 47
EL.U/mL
  Anti-PD, Month 0: number analyzed (Participants) | 47 | 46
  Anti-PD, Month 0 | 79.59 [62.08 to 102.04] | 76.22 [61.39 to 94.63]
  Anti-PD, Month 2 | 199.23 [150.51 to 263.72] | 184.34 [140.21 to 242.35]
  Anti-PD, Month 3: number analyzed (Participants) | 48 | 46
  Anti-PD, Month 3 | 1376.56 [1020.71 to 1856.46] | 760.99 [553.23 to 1046.77]

12. Secondary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes for Subjects Receiving Synflorix Vaccine Co-administered With Tritanrix-HepB/Hib and Polio Sabin Vaccines
Description: Opsonophagocytic activity has been assessed against vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (OPA-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) and presented as geometric mean titers (GMTs). The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: as for outcome 6
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who were co-administered Synflorix with Tritanrix-HepB/Hib and Polio Sabin vaccines, for whom opsonophagocytic activity assay results for antibodies against at least one vaccine antigen component were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 46 | 41
Titer
  OPA-1, Month 3: number analyzed (Participants) | 45 | 41
  OPA-1, Month 3 | 106.4 [56.0 to 202.2] | 94.6 [49.9 to 179.5]
  OPA-1, Month 8: number analyzed (Participants) | 41 | 33
  OPA-1, Month 8 | 11.7 [6.8 to 20.1] | 10.9 [6.0 to 20.1]
  OPA-1, Month 9: number analyzed (Participants) | 41 | 35
  OPA-1, Month 9 | 930.5 [606.3 to 1427.9] | 750.4 [401.4 to 1403.0]
  OPA-4, Month 3: number analyzed (Participants) | 44 | 38
  OPA-4, Month 3 | 1316.6 [1014.0 to 1709.7] | 992.5 [680.0 to 1448.4]
  OPA-4, Month 8: number analyzed (Participants) | 40 | 31
  OPA-4, Month 8 | 222.1 [130.6 to 377.8] | 108.3 [51.6 to 227.6]
  OPA-4, Month 9: number analyzed (Participants) | 41 | 33
  OPA-4, Month 9 | 2064.2 [1625.3 to 2621.8] | 2079.3 [1425.7 to 3032.7]
  OPA-5, Month 3: number analyzed (Participants) | 44 | 41
  OPA-5, Month 3 | 106.9 [66.8 to 171.2] | 119.4 [81.4 to 175.2]
  OPA-5, Month 8: number analyzed (Participants) | 40 | 33
  OPA-5, Month 8 | 14.9 [8.9 to 24.9] | 15.8 [9.6 to 26.1]
  OPA-5, Month 9: number analyzed (Participants) | 41 | 33
  OPA-5, Month 9 | 273.2 [200.6 to 372.0] | 277.5 [168.8 to 456.1]
  OPA-6B, Month 3: number analyzed (Participants) | 41 | 37
  OPA-6B, Month 3 | 1043.3 [605.3 to 1798.3] | 446.2 [207.4 to 960.0]
  OPA-6B, Month 8: number analyzed (Participants) | 39 | 32
  OPA-6B, Month 8 | 285.3 [150.1 to 542.1] | 245.6 [115.0 to 524.3]
  OPA-6B, Month 9: number analyzed (Participants) | 40 | 33
  OPA-6B, Month 9 | 952.2 [638.8 to 1419.3] | 989.2 [530.6 to 1843.9]
  OPA-7F, Month 3: number analyzed (Participants) | 42 | 37
  OPA-7F, Month 3 | 4644.1 [3519.3 to 6128.4] | 4924.2 [3430.2 to 7068.8]
  OPA-7F, Month 8: number analyzed (Participants) | 40 | 32
  OPA-7F, Month 8 | 1747.2 [1225.4 to 2491.3] | 1585.7 [1133.8 to 2217.8]
  OPA-7F, Month 9: number analyzed (Participants) | 39 | 32
  OPA-7F, Month 9 | 7262.9 [5257.6 to 10033.1] | 8120.3 [5802.1 to 11364.8]
  OPA-9V, Month 3: number analyzed (Participants) | 46 | 39
  OPA-9V, Month 3 | 1438.6 [1084.0 to 1909.3] | 1116.8 [679.6 to 1835.2]
  OPA-9V, Month 8: number analyzed (Participants) | 38 | 32
  OPA-9V, Month 8 | 215.5 [97.5 to 476.1] | 244.5 [123.9 to 482.2]
  OPA-9V, Month 9: number analyzed (Participants) | 40 | 32
  OPA-9V, Month 9 | 2062.3 [1569.0 to 2710.8] | 2987.2 [2149.4 to 4151.6]
  OPA-14, Month 3: number analyzed (Participants) | 44 | 41
  OPA-14, Month 3 | 1689.9 [1090.7 to 2618.2] | 1062.3 [562.8 to 2005.2]
  OPA-14, Month 8: number analyzed (Participants) | 39 | 26
  OPA-14, Month 8 | 215.9 [113.6 to 410.1] | 132.5 [60.3 to 291.5]
  OPA-14, Month 9: number analyzed (Participants) | 40 | 33
  OPA-14, Month 9 | 1571.5 [1114.2 to 2216.4] | 1454.1 [741.8 to 2850.5]
  OPA-18C, Month 3: number analyzed (Participants) | 40 | 37
  OPA-18C, Month 3 | 873.8 [591.7 to 1290.4] | 524.7 [319.6 to 861.6]
  OPA-18C, Month 8: number analyzed (Participants) | 39 | 30
  OPA-18C, Month 8 | 46.5 [28.5 to 75.7] | 28.7 [17.5 to 47.3]
  OPA-18C, Month 9: number analyzed (Participants) | 39 | 31
  OPA-18C, Month 9 | 1246.0 [776.7 to 1999.0] | 1011.8 [686.4 to 1491.4]
  OPA-19F, Month 3: number analyzed (Participants) | 43 | 39
  OPA-19F, Month 3 | 558.9 [376.3 to 830.2] | 266.1 [148.2 to 477.8]
  OPA-19F, Month 8: number analyzed (Participants) | 41 | 32
  OPA-19F, Month 8 | 60.7 [37.1 to 99.3] | 43.4 [22.6 to 83.2]
  OPA-19F, Month 9: number analyzed (Participants) | 40 | 33
  OPA-19F, Month 9 | 652.9 [413.3 to 1031.5] | 486.7 [278.9 to 849.4]
  OPA-23F, Month 3: number analyzed (Participants) | 44 | 37
  OPA-23F, Month 3 | 705.1 [309.2 to 1607.8] | 759.7 [326.7 to 1766.6]
  OPA-23F, Month 8: number analyzed (Participants) | 36 | 31
  OPA-23F, Month 8 | 85.2 [27.5 to 264.4] | 41.6 [14.6 to 118.9]
  OPA-23F, Month 9: number analyzed (Participants) | 39 | 33
  OPA-23F, Month 9 | 4231.2 [2793.7 to 6408.3] | 1454.0 [736.1 to 2872.3]

13. Secondary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes for Subjects Who Received a Two-dose Primary Vaccination Followed by a Booster Dose
Description: as for outcome 12
Time Frame: as for outcome 4
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose primary vaccination followed by a booster dose, for whom opsonophagocytic activity assay results for antibodies against at least one vaccine antigen component were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 7-11S Group | Synflorix 7-11NS Group
Number analyzed (Participants) | 49 | 47
Titer
  OPA-1, Month 0: number analyzed (Participants) | 47 | 43
  OPA-1, Month 0 | 4.9 [3.8 to 6.3] | 4.5 [3.6 to 5.7]
  OPA-1, Month 2: number analyzed (Participants) | 48 | 45
  OPA-1, Month 2 | 134.7 [83.6 to 216.9] | 88.1 [53.7 to 144.6]
  OPA-1, Month 3: number analyzed (Participants) | 48 | 46
  OPA-1, Month 3 | 74.2 [42.6 to 129.3] | 48.0 [26.6 to 86.7]
  OPA-1, Month 4: number analyzed (Participants) | 48 | 44
  OPA-1, Month 4 | 516.0 [307.6 to 865.7] | 511.3 [293.2 to 891.8]
  OPA-4, Month 0: number analyzed (Participants) | 44 | 44
  OPA-4, Month 0 | 5.1 [3.6 to 7.2] | 11.8 [5.7 to 24.5]
  OPA-4, Month 2: number analyzed (Participants) | 49 | 44
  OPA-4, Month 2 | 1636.3 [1217.5 to 2199.2] | 1771.1 [1359.0 to 2308.2]
  OPA-4, Month 3: number analyzed (Participants) | 45 | 45
  OPA-4, Month 3 | 812.7 [584.5 to 1130.1] | 1048.3 [790.4 to 1390.3]
  OPA-4, Month 4: number analyzed (Participants) | 48 | 43
  OPA-4, Month 4 | 2130.5 [1639.1 to 2769.2] | 2415.5 [1686.5 to 3459.8]
  OPA-5, Month 0: number analyzed (Participants) | 47 | 44
  OPA-5, Month 0 | 4.4 [3.8 to 5.1] | 4.0 [4.0 to 4.0]
  OPA-5, Month 2: number analyzed (Participants) | 49 | 46
  OPA-5, Month 2 | 105.7 [67.7 to 165.1] | 85.8 [59.4 to 124.0]
  OPA-5, Month 3: number analyzed (Participants) | 47 | 47
  OPA-5, Month 3 | 54.1 [34.9 to 83.6] | 49.2 [31.7 to 76.3]
  OPA-5, Month 4: number analyzed (Participants) | 48 | 43
  OPA-5, Month 4 | 277.4 [180.7 to 425.7] | 289.6 [190.9 to 439.3]
  OPA-6B, Month 0: number analyzed (Participants) | 43 | 41
  OPA-6B, Month 0 | 7.9 [4.6 to 13.8] | 8.5 [4.7 to 15.4]
  OPA-6B, Month 2: number analyzed (Participants) | 48 | 43
  OPA-6B, Month 2 | 702.5 [413.2 to 1194.2] | 696.6 [388.5 to 1249.2]
  OPA-6B, Month 3: number analyzed (Participants) | 44 | 45
  OPA-6B, Month 3 | 708.3 [422.9 to 1186.1] | 615.5 [337.3 to 1123.1]
  OPA-6B, Month 4: number analyzed (Participants) | 46 | 43
  OPA-6B, Month 4 | 1360.0 [860.2 to 2150.3] | 1305.4 [731.9 to 2328.4]
  OPA-7F, Month 0: number analyzed (Participants) | 41 | 40
  OPA-7F, Month 0 | 215.3 [91.2 to 508.1] | 643.5 [293.4 to 1411.7]
  OPA-7F, Month 2: number analyzed (Participants) | 47 | 40
  OPA-7F, Month 2 | 6694.3 [5055.1 to 8864.9] | 10452.0 [7782.7 to 14036.6]
  OPA-7F, Month 3: number analyzed (Participants) | 46 | 46
  OPA-7F, Month 3 | 7776.9 [6000.8 to 10078.7] | 9336.3 [6752.4 to 12908.9]
  OPA-7F, Month 4: number analyzed (Participants) | 47 | 39
  OPA-7F, Month 4 | 10854.8 [9051.6 to 13017.2] | 9362.8 [6882.3 to 12737.3]
  OPA-9V, Month 0: number analyzed (Participants) | 42 | 44
  OPA-9V, Month 0 | 16.9 [8.3 to 34.5] | 20.3 [9.2 to 44.5]
  OPA-9V, Month 2: number analyzed (Participants) | 48 | 42
  OPA-9V, Month 2 | 2858.2 [1875.3 to 4356.2] | 2667.9 [1677.9 to 4242.0]
  OPA-9V, Month 3: number analyzed (Participants) | 44 | 46
  OPA-9V, Month 3 | 1982.9 [1192.1 to 3298.2] | 1986.2 [1167.8 to 3378.2]
  OPA-9V, Month 4: number analyzed (Participants) | 48 | 41
  OPA-9V, Month 4 | 3047.9 [2389.7 to 3887.3] | 2719.2 [1681.0 to 4398.9]
  OPA-14, Month 0: number analyzed (Participants) | 40 | 39
  OPA-14, Month 0 | 5.5 [3.8 to 8.1] | 5.9 [3.8 to 9.1]
  OPA-14, Month 2: number analyzed (Participants) | 44 | 43
  OPA-14, Month 2 | 2109.5 [1299.0 to 3425.9] | 4009.9 [2501.9 to 6426.7]
  OPA-14, Month 3: number analyzed (Participants) | 46 | 46
  OPA-14, Month 3 | 1431.6 [865.2 to 2368.6] | 2128.3 [1477.5 to 3065.9]
  OPA-14, Month 4: number analyzed (Participants) | 46 | 40
  OPA-14, Month 4 | 3414.9 [2237.4 to 5211.9] | 3717.3 [2403.9 to 5748.5]
  OPA-18C, Month 0: number analyzed (Participants) | 44 | 43
  OPA-18C, Month 0 | 4.1 [3.9 to 4.5] | 4.6 [3.4 to 6.2]
  OPA-18C, Month 2: number analyzed (Participants) | 39 | 37
  OPA-18C, Month 2 | 744.4 [393.3 to 1409.2] | 1605.6 [937.1 to 2751.1]
  OPA-18C, Month 3: number analyzed (Participants) | 40 | 42
  OPA-18C, Month 3 | 411.4 [214.4 to 789.7] | 746.4 [430.5 to 1294.1]
  OPA-18C, Month 4: number analyzed (Participants) | 44 | 40
  OPA-18C, Month 4 | 2218.9 [1577.5 to 3121.2] | 3238.7 [1874.7 to 5595.0]
  OPA-19F, Month 0: number analyzed (Participants) | 44 | 43
  OPA-19F, Month 0 | 4.2 [3.8 to 4.7] | 4.0 [4.0 to 4.0]
  OPA-19F, Month 2: number analyzed (Participants) | 47 | 43
  OPA-19F, Month 2 | 393.4 [214.4 to 722.0] | 491.5 [256.8 to 940.6]
  OPA-19F, Month 3: number analyzed (Participants) | 45 | 46
  OPA-19F, Month 3 | 160.2 [86.8 to 295.6] | 279.5 [161.1 to 484.9]
  OPA-19F, Month 4: number analyzed (Participants) | 47 | 41
  OPA-19F, Month 4 | 1347.7 [813.6 to 2232.3] | 1174.4 [605.6 to 2277.3]
  OPA-23F, Month 0: number analyzed (Participants) | 43 | 40
  OPA-23F, Month 0 | 7.6 [4.1 to 13.9] | 15.3 [6.4 to 36.6]
  OPA-23F, Month 2: number analyzed (Participants) | 46 | 44
  OPA-23F, Month 2 | 1545.1 [788.3 to 3028.2] | 2107.5 [1155.0 to 3845.5]
  OPA-23F, Month 3: number analyzed (Participants) | 40 | 46
  OPA-23F, Month 3 | 1168.8 [560.8 to 2435.8] | 1026.2 [458.3 to 2298.0]
  OPA-23F, Month 4: number analyzed (Participants) | 47 | 43
  OPA-23F, Month 4 | 2038.8 [977.1 to 4254.4] | 3525.1 [1974.2 to 6294.4]

14. Secondary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes for Subjects Who Received a Two-dose Primary Vaccination Without Any Booster Dose
Description: as for outcome 12
Time Frame: Prior to (Month 0) the first vaccine dose, prior to (Month 2) and one month after (Month 3) the second vaccine dose
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose vaccination without any booster dose, for whom data concerning immunogenicity outcomes and opsonophagocytic activity assay results for antibodies against at least one vaccine antigen component were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 47 | 45
Titer
  OPA-1, Month 0: number analyzed (Participants) | 47 | 43
  OPA-1, Month 0 | 6.9 [4.5 to 10.8] | 5.6 [4.2 to 7.6]
  OPA-1, Month 2: number analyzed (Participants) | 46 | 45
  OPA-1, Month 2 | 9.3 [6.1 to 14.3] | 10.9 [6.8 to 17.4]
  OPA-1, Month 3: number analyzed (Participants) | 45 | 43
  OPA-1, Month 3 | 195.7 [119.9 to 319.3] | 115.1 [64.0 to 206.8]
  OPA-4, Month 0: number analyzed (Participants) | 46 | 44
  OPA-4, Month 0 | 8.0 [4.7 to 13.6] | 7.3 [4.3 to 12.3]
  OPA-4, Month 2: number analyzed (Participants) | 44 | 43
  OPA-4, Month 2 | 1086.3 [758.4 to 1555.9] | 1539.4 [1128.4 to 2100.1]
  OPA-4, Month 3: number analyzed (Participants) | 44 | 43
  OPA-4, Month 3 | 2089.7 [1635.0 to 2670.8] | 3193.9 [2241.3 to 4551.4]
  OPA-5, Month 0 | 5.5 [4.2 to 7.4] | 4.4 [3.6 to 5.4]
  OPA-5, Month 2: number analyzed (Participants) | 45 | 45
  OPA-5, Month 2 | 9.8 [7.1 to 13.7] | 9.6 [6.6 to 13.7]
  OPA-5, Month 3: number analyzed (Participants) | 44 | 44
  OPA-5, Month 3 | 151.3 [99.8 to 229.2] | 84.0 [53.5 to 131.8]
  OPA-6B, Month 0: number analyzed (Participants) | 41 | 38
  OPA-6B, Month 0 | 13.6 [6.7 to 27.6] | 9.9 [5.2 to 18.7]
  OPA-6B, Month 2: number analyzed (Participants) | 41 | 42
  OPA-6B, Month 2 | 345.1 [172.4 to 690.7] | 278.4 [131.8 to 588.4]
  OPA-6B, Month 3: number analyzed (Participants) | 43 | 43
  OPA-6B, Month 3 | 748.4 [425.9 to 1315.0] | 866.4 [511.8 to 1466.7]
  OPA-7F, Month 0: number analyzed (Participants) | 44 | 36
  OPA-7F, Month 0 | 1436.6 [1014.4 to 2034.6] | 1228.1 [783.3 to 1925.5]
  OPA-7F, Month 2: number analyzed (Participants) | 44 | 45
  OPA-7F, Month 2 | 5462.3 [4108.9 to 7261.4] | 5802.2 [4678.6 to 7195.6]
  OPA-7F, Month 3: number analyzed (Participants) | 44 | 42
  OPA-7F, Month 3 | 10279.4 [7836.7 to 13483.6] | 10131.4 [8303.7 to 12361.6]
  OPA-9V, Month 0: number analyzed (Participants) | 40 | 37
  OPA-9V, Month 0 | 119.5 [50.4 to 283.2] | 81.3 [35.7 to 185.0]
  OPA-9V, Month 2: number analyzed (Participants) | 43 | 44
  OPA-9V, Month 2 | 1976.2 [1392.6 to 2804.4] | 2359.0 [1514.3 to 3674.9]
  OPA-9V, Month 3: number analyzed (Participants) | 44 | 43
  OPA-9V, Month 3 | 3778.2 [2880.0 to 4956.4] | 4276.8 [3122.3 to 5858.3]
  OPA-14, Month 0: number analyzed (Participants) | 40 | 34
  OPA-14, Month 0 | 16.3 [8.3 to 31.8] | 12.0 [5.3 to 27.0]
  OPA-14, Month 2: number analyzed (Participants) | 42 | 40
  OPA-14, Month 2 | 711.2 [400.7 to 1262.4] | 865.6 [583.2 to 1284.9]
  OPA-14, Month 3: number analyzed (Participants) | 45 | 40
  OPA-14, Month 3 | 2704.5 [1856.4 to 3940.0] | 2737.5 [1890.0 to 3965.1]
  OPA-18C, Month 0: number analyzed (Participants) | 44 | 40
  OPA-18C, Month 0 | 4.9 [4.0 to 6.0] | 4.0 [4.0 to 4.0]
  OPA-18C, Month 2: number analyzed (Participants) | 32 | 34
  OPA-18C, Month 2 | 1035.5 [507.6 to 2112.5] | 449.2 [222.8 to 905.9]
  OPA-18C, Month 3: number analyzed (Participants) | 40 | 40
  OPA-18C, Month 3 | 2873.1 [2070.0 to 3987.6] | 2126.8 [1509.7 to 2996.3]
  OPA-19F, Month 0: number analyzed (Participants) | 46 | 42
  OPA-19F, Month 0 | 5.5 [4.2 to 7.3] | 4.0 [4.0 to 4.0]
  OPA-19F, Month 2: number analyzed (Participants) | 44 | 43
  OPA-19F, Month 2 | 229.1 [132.9 to 395.0] | 248.0 [143.0 to 430.1]
  OPA-19F, Month 3: number analyzed (Participants) | 45 | 43
  OPA-19F, Month 3 | 1845.3 [1169.3 to 2912.1] | 1271.4 [825.4 to 1958.3]
  OPA-23F, Month 0: number analyzed (Participants) | 39 | 38
  OPA-23F, Month 0 | 68.1 [21.1 to 219.6] | 37.6 [12.3 to 114.3]
  OPA-23F, Month 2: number analyzed (Participants) | 44 | 44
  OPA-23F, Month 2 | 2572.2 [1264.1 to 5233.9] | 2433.6 [1309.7 to 4522.0]
  OPA-23F, Month 3: number analyzed (Participants) | 42 | 41
  OPA-23F, Month 3 | 5016.6 [3176.6 to 7922.4] | 5325.4 [2857.8 to 9923.9]

15. Secondary Outcome: Opsonophagocytic Titers Against Cross-reactive Pneumococcal Serotypes for Subjects Receiving Synflorix Vaccine Co-administered With Tritanrix-HepB/Hib and Polio Sabin Vaccines
Description: Opsonophagocytic activity has been assessed for cross-reactive vaccine pneumococcal serotypes 6A and 19A (OPA-6A, OPA-19A) and presented as geometric mean titers (GMTs). The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: as for outcome 6
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who were co-administered Synflorix with Tritanrix-HepB/Hib and Polio Sabin vaccines, for whom opsonophagocytic activity assay results for antibodies against at least one cross-reactive pneumococcal serotype were available for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 42 | 41
Titer
  OPA-6A, Month 3 | 24.73 [11.46 to 53.37] | 9.45 [5.32 to 16.75]
  OPA-6A, Month 8: number analyzed (Participants) | 40 | 33
  OPA-6A, Month 8 | 18.23 [8.97 to 37.09] | 17.59 [8.08 to 38.30]
  OPA-6A, Month 9: number analyzed (Participants) | 38 | 32
  OPA-6A, Month 9 | 35.35 [15.60 to 80.12] | 30.70 [12.14 to 77.64]
  OPA-19A, Month 3: number analyzed (Participants) | 38 | 34
  OPA-19A, Month 3 | 9.42 [5.65 to 15.70] | 5.04 [3.83 to 6.63]
  OPA-19A, Month 8: number analyzed (Participants) | 34 | 23
  OPA-19A, Month 8 | 6.31 [4.28 to 9.32] | 5.83 [3.95 to 8.61]
  OPA-19A, Month 9: number analyzed (Participants) | 26 | 28
  OPA-19A, Month 9 | 22.06 [9.49 to 51.30] | 19.44 [10.25 to 36.86]

16. Secondary Outcome: Opsonophagocytic Titers Against Cross-reactive Pneumococcal Serotypes for Subjects Who Received a Two-dose Primary Vaccination Followed by a Booster Dose
Description: as for outcome 15
Time Frame: as for outcome 4
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose primary vaccination followed by a booster dose, for whom opsonophagocytic activity assay results for antibodies against at least one cross-reactive pneumococcal serotype were available for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 7-11S Group | Synflorix 7-11NS Group
Number analyzed (Participants) | 49 | 45
Titer
  OPA-6A, Month 0: number analyzed (Participants) | 46 | 40
  OPA-6A, Month 0 | 4.81 [3.71 to 6.24] | 5.02 [3.64 to 6.90]
  OPA-6A, Month 2: number analyzed (Participants) | 49 | 39
  OPA-6A, Month 2 | 40.59 [19.11 to 86.23] | 51.23 [22.85 to 114.88]
  OPA-6A, Month 3: number analyzed (Participants) | 44 | 45
  OPA-6A, Month 3 | 38.11 [17.04 to 85.21] | 36.27 [16.89 to 77.89]
  OPA-6A, Month 4: number analyzed (Participants) | 45 | 43
  OPA-6A, Month 4 | 77.09 [35.58 to 167.04] | 98.18 [43.05 to 223.96]
  OPA-19A, Month 0: number analyzed (Participants) | 41 | 40
  OPA-19A, Month 0 | 4.49 [3.91 to 5.16] | 4.33 [3.68 to 5.10]
  OPA-19A, Month 2: number analyzed (Participants) | 40 | 31
  OPA-19A, Month 2 | 15.21 [7.95 to 29.08] | 108.31 [49.55 to 236.78]
  OPA-19A, Month 3: number analyzed (Participants) | 37 | 26
  OPA-19A, Month 3 | 14.65 [7.71 to 27.81] | 19.40 [8.04 to 46.82]
  OPA-19A, Month 4: number analyzed (Participants) | 31 | 29
  OPA-19A, Month 4 | 76.09 [30.50 to 189.83] | 449.06 [170.05 to 1185.87]

17. Secondary Outcome: Opsonophagocytic Titers Against Cross-reactive Pneumococcal Serotypes for Subjects Who Received a Two-dose Primary Vaccination Without Any Booster Dose
Description: as for outcome 15
Time Frame: Prior to (Month 0) the first vaccine dose, prior to (Month 2) and one month after (Month 3) the second vaccine dose
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who received a two-dose vaccination without any booster dose, for whom opsonophagocytic activity assay results for antibodies against at least one cross-reactive pneumococcal serotype were available for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 44 | 42
Titer
  OPA-6A, Month 0: number analyzed (Participants) | 44 | 40
  OPA-6A, Month 0 | 9.26 [5.76 to 14.89] | 6.35 [4.02 to 10.02]
  OPA-6A, Month 2 | 82.82 [40.27 to 170.33] | 77.25 [31.81 to 187.64]
  OPA-6A, Month 3: number analyzed (Participants) | 40 | 39
  OPA-6A, Month 3 | 147.91 [63.11 to 346.68] | 157.37 [59.23 to 418.11]
  OPA-19A, Month 0: number analyzed (Participants) | 44 | 40
  OPA-19A, Month 0 | 5.85 [4.27 to 8.01] | 6.32 [4.09 to 9.76]
  OPA-19A, Month 2: number analyzed (Participants) | 23 | 27
  OPA-19A, Month 2 | 28.37 [11.84 to 67.98] | 25.68 [11.60 to 56.84]
  OPA-19A, Month 3: number analyzed (Participants) | 19 | 23
  OPA-19A, Month 3 | 214.17 [75.58 to 606.93] | 321.14 [144.75 to 712.50]

18. Secondary Outcome: Concentration of Antibodies Against Diphtheria Toxoid (DT) and Tetanus Toxoid (TT) for Subjects Who Were Co-administered Tritanrix-HepB/Hib Vaccine
Description: Anti-DT and anti-TT antibody concentrations are presented as geometric mean concentrations (GMCs) and expressed in international units per milliliter (IU/mL). Seroprotection status was defined as anti-DT or anti-TT antibody concentration ≥ than 0.1 IU/mL.
Time Frame: as for outcome 6
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who were co-administered Tritanrix-HepB/Hib vaccine, for whom data concerning immunogenicity outcomes and assay results for antibodies against diphtheria and tetanus toxoids were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 48 | 46
IU/mL
  Anti-DT, Month 0: number analyzed (Participants) | 48 | 45
  Anti-DT, Month 0 | 0.07 [0.05 to 0.08] | 0.06 [0.05 to 0.07]
  Anti-DT, Month 3 | 3.22 [2.59 to 4.00] | 3.50 [2.82 to 4.34]
  Anti-DT, Month 8: number analyzed (Participants) | 44 | 37
  Anti-DT, Month 8 | 0.62 [0.50 to 0.77] | 0.90 [0.72 to 1.12]
  Anti-DT, Month 9: number analyzed (Participants) | 44 | 38
  Anti-DT, Month 9 | 6.58 [5.44 to 7.97] | 7.55 [6.11 to 9.32]
  Anti-TT, Month 0 | 1.54 [1.13 to 2.09] | 1.22 [0.85 to 1.76]
  Anti-TT, Month 3 | 4.04 [3.26 to 5.01] | 4.13 [3.27 to 5.22]
  Anti-TT, Month 8: number analyzed (Participants) | 44 | 38
  Anti-TT, Month 8 | 1.19 [0.96 to 1.48] | 1.33 [1.08 to 1.63]
  Anti-TT, Month 9: number analyzed (Participants) | 44 | 38
  Anti-TT, Month 9 | 10.88 [9.24 to 12.81] | 11.11 [9.62 to 12.83]

19. Secondary Outcome: Concentrations of Antibodies Against Bordetella Pertussis (BPT) for Subjects Who Were Co-administered Tritanrix-HepB/Hib Vaccine
Description: Anti-BPT antibody concentrations are presented as geometric mean concentrations (GMCs) and expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 15 EL.U/mL.
Time Frame: as for outcome 6
Population: The analysis was performed on the ATP immunogenicity cohort and included all subjects who were co-administered Tritanrix-HepB/Hib vaccine, for whom data concerning immunogenicity outcomes and assay results for antibodies against Bordetella pertussis were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group
Number analyzed (Participants) | 48 | 46
EL.U/mL
  Anti-BPT, Month 0 | 7.71 [7.29 to 8.16] | 7.77 [7.39 to 8.17]
  Anti-BPT, Month 3 | 105.61 [86.93 to 128.30] | 101.74 [84.56 to 122.42]
  Anti-BPT, Month 8: number analyzed (Participants) | 44 | 38
  Anti-BPT, Month 8 | 22.67 [17.45 to 29.45] | 22.69 [17.88 to 28.80]
  Anti-BPT, Month 9: number analyzed (Participants) | 44 | 38
  Anti-BPT, Month 9 | 177.87 [152.10 to 207.99] | 190.58 [167.67 to 216.63]

20. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms During the Primary Vaccination Phase
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-primary vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort for the primary epoch, which included all vaccinated subjects who completed their symptoms sheet for the respective dose. Note that dose 3 rows are not applicable for subjects from the 7-11 and 12-23 months of age groups as they only received a 2-dose primary vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50
Participants
  Any Pain, Dose 1 | 8 | 12 | 7 | 10 | 9 | 6
  Grade 3 Pain, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Any Pain, Dose 2 | 7 | 7 | 5 | 7 | 5 | 3
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Grade 3 Pain, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Any Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Any Swelling, Dose 2 | 0 | 1 | 0 | 1 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Any Pain, Dose 3 | 4 | 6 |  |  |  |
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Grade 3 Pain, Dose 3 | 0 | 0 |  |  |  |
  Any Redness, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Any Redness, Dose 3 | 0 | 0 |  |  |  |
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Grade 3 Redness, Dose 3 | 0 | 0 |  |  |  |
  Any Swelling, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Any Swelling, Dose 3 | 0 | 0 |  |  |  |
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Grade 3 Swelling, Dose 3 | 0 | 0 |  |  |  |
  Any Pain, Across doses | 17 | 23 | 12 | 15 | 13 | 9
  Grade 3 Pain, Across doses | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness, Across doses | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Redness, Across doses | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Across doses | 0 | 1 | 0 | 1 | 1 | 1
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms During the Booster Vaccination Phase
Description: as for outcome 20
Time Frame: During the 4-day (Days 0-3) post-booster vaccination period
Population: The analysis was performed on the Total Vaccinated cohort for the booster epoch, which included all booster vaccinated subjects who completed their symptoms sheet. Note that no data are reported for the 12-23 months of age groups as they were not administered any vaccine during the booster phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 49 | 49 | 50 | 50 | 0 | 0
Participants
  Any Pain | 11 | 6 | 3 | 0 |  |
  Grade 3 Pain | 0 | 0 | 0 | 0 |  |
  Any Redness | 0 | 0 | 0 | 0 |  |
  Grade 3 Redness | 0 | 0 | 0 | 0 |  |
  Any Swelling | 1 | 0 | 1 | 0 |  |
  Grade 3 Swelling | 0 | 0 | 0 | 0 |  |

22. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms During the Primary Vaccination Phase
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as rectal temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 40.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-primary vaccination period following each dose and across doses
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50
Participants
  Any Drowsiness, Dose 1 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Drowsiness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 1 | 0 | 0 | 0 | 1 | 0 | 0
  Any Irritability, Dose 1 | 0 | 2 | 0 | 0 | 1 | 0
  Grade 3 Irritability, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Irritability, Dose 1 | 0 | 0 | 0 | 0 | 1 | 0
  Any Loss of appetite, Dose 1 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Loss of appetite, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Loss of appetite, Dose 1 | 0 | 0 | 0 | 0 | 0 | 1
  Any Fever, Dose 1 | 34 | 31 | 22 | 26 | 21 | 15
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 31 | 29 | 19 | 22 | 21 | 13
  Any Drowsiness, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Any Drowsiness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Grade 3 Drowsiness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Related Drowsiness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Any Irritability, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Any Irritability, Dose 2 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Grade 3 Irritability, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Related Irritability, Dose 2 | 0 | 0 | 0 | 0 | 1 | 0
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Any Loss of appetite, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Grade 3 Loss of appetite, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Related Loss of appetite, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Any Fever, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Any Fever, Dose 2 | 40 | 30 | 22 | 11 | 12 | 12
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Grade 3 Fever, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 48
  Related Fever, Dose 2 | 38 | 28 | 20 | 9 | 10 | 9
  Any Drowsiness, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Any Drowsiness, Dose 3 | 0 | 0 |  |  |  |
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 3 | 0 | 0 |  |  |  |
  Related Drowsiness, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 3 | 0 | 0 |  |  |  |
  Any Irritability, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Any Irritability, Dose 3 | 3 | 4 |  |  |  |
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Grade 3 Irritability, Dose 3 | 0 | 0 |  |  |  |
  Related Irritability, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Related Irritability, Dose 3 | 3 | 3 |  |  |  |
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Any Loss of appetite, Dose 3 | 0 | 1 |  |  |  |
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Grade 3 Loss of appetite, Dose 3 | 0 | 0 |  |  |  |
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Related Loss of appetite, Dose 3 | 0 | 0 |  |  |  |
  Any Fever, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Any Fever, Dose 3 | 30 | 30 |  |  |  |
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Grade 3 Fever, Dose 3 | 0 | 0 |  |  |  |
  Related Fever, Dose 3: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0 | 0
  Related Fever, Dose 3 | 26 | 28 |  |  |  |
  Any Drowsiness, Across doses | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Drowsiness, Across doses | 0 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Across doses | 0 | 0 | 0 | 1 | 0 | 0
  Any Irritability, Across doses | 3 | 6 | 0 | 0 | 2 | 0
  Grade 3 Irritability, Across doses | 0 | 0 | 0 | 0 | 0 | 0
  Related Irritability, Across doses | 3 | 3 | 0 | 0 | 2 | 0
  Any Loss of appetite, Across doses | 0 | 1 | 0 | 0 | 0 | 1
  Grade 3 Loss of appetite, Across doses | 0 | 0 | 0 | 0 | 0 | 0
  Related Loss of appetite, Across doses | 0 | 0 | 0 | 0 | 0 | 1
  Any Fever, Across doses | 48 | 43 | 31 | 29 | 29 | 20
  Grade 3 Fever, Across doses | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Across doses | 46 | 43 | 29 | 25 | 28 | 17

23. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms During the Booster Vaccination Phase
Description: as for outcome 22
Time Frame: During the 4-day (Days 0-3) post-booster vaccination period
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 49 | 49 | 50 | 50 | 0 | 0
Participants
  Any Drowsiness | 0 | 0 | 0 | 0 |  |
  Grade 3 Drowsiness | 0 | 0 | 0 | 0 |  |
  Related Drowsiness | 0 | 0 | 0 | 0 |  |
  Any Irritability | 6 | 0 | 0 | 0 |  |
  Grade 3 Irritability | 0 | 0 | 0 | 0 |  |
  Related Irritability | 5 | 0 | 0 | 0 |  |
  Any Loss of appetite | 0 | 0 | 0 | 0 |  |
  Grade 3 Loss of appetite | 0 | 0 | 0 | 0 |  |
  Related Loss of appetite | 0 | 0 | 0 | 0 |  |
  Any Fever | 38 | 31 | 14 | 13 |  |
  Grade 3 Fever | 0 | 0 | 0 | 0 |  |
  Related Fever | 35 | 28 | 13 | 13 |  |

24. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 31-day (Days 0-30) post-primary and post-booster vaccination period
Population: The analysis was performed on the Total Vaccinated cohort for the primary and booster epochs, which included all vaccinated subjects who received at least one dose of primary vaccination and the booster dose of study vaccine, respectively. Note that subjects from the 12-23 months of age groups did not participate in the Booster Epoch.
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50
Participants
  Any AE(s), post-primary vaccination | 37 | 34 | 32 | 37 | 23 | 25
  Any AE(s), post-booster vaccination: number analyzed (Participants) | 49 | 49 | 50 | 50 | 0 | 0
  Any AE(s), post-booster vaccination | 8 | 17 | 18 | 12 |  |

25. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period from Month 0 to Month 9
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who received at least one dose of vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50
Participants | 3 | 9 | 3 | 4 | 2 | 2

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) period following each vaccination dose; Unsolicited AEs: within the 31-day (Days 0-30) period following each vaccination; SAEs: throughout the study, from Day 0 up to Month 9.
Arm/Group | Tritanrix-HepB/Hib+Polio Sabin <6S Group | Tritanrix-HepB/Hib+Polio Sabin <6NS Group | Synflorix 7-11S Group | Synflorix 7-11NS Group | Synflorix 12-23S Group | Synflorix 12-23NS Group
All-Cause Mortality (participants affected / at risk) | 1/50 | 1/50 | 1/50 | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 9/50 | 3/50 | 4/50 | 2/50 | 2/50
Other Adverse Events (participants affected / at risk) | 50/50 | 49/50 | 47/50 | 47/50 | 41/50 | 31/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tritanrix-HepB/Hib+Polio Sabin <6S Group (N=50) | Tritanrix-HepB/Hib+Polio Sabin <6NS Group (N=50) | Synflorix 7-11S Group (N=50) | Synflorix 7-11NS Group (N=50) | Synflorix 12-23S Group (N=50) | Synflorix 12-23NS Group (N=50)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Meningitis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tritanrix-HepB/Hib+Polio Sabin <6S Group (N=50) | Tritanrix-HepB/Hib+Polio Sabin <6NS Group (N=50) | Synflorix 7-11S Group (N=50) | Synflorix 7-11NS Group (N=50) | Synflorix 12-23S Group (N=50) | Synflorix 12-23NS Group (N=50)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 9 (10) | 10 (12) | 6 (6) | 9 (10) | 1 (1) | 4 (4)
Conjunctivitis (Eye disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 6 (6) | 4 (4) | 4 (4) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 2 (2) | 5 (5) | 7 (7) | 4 (4) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (6) | 6 (7) | 3 (3) | 7 (7) | 1 (1) | 5 (5)
Gastrointestinal fungal infection (Infections and infestations) | 4 (5) | 6 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 9 (9) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaria (Infections and infestations) | 10 (10) | 13 (14) | 18 (19) | 18 (20) | 10 (10) | 8 (8)
Nasopharyngitis (Infections and infestations) | 7 (7) | 5 (6) | 3 (3) | 8 (8) | 4 (4) | 5 (5)
Pain (General disorders) | 23 (30) | 26 (31) | 15 (17) | 15 (17) | 14 (16) | 9 (9)
Pyrexia (General disorders) | 49 (143) | 47 (123) | 37 (63) | 35 (52) | 29 (33) | 21 (28)
Rhinitis (Infections and infestations) | 4 (4) | 7 (7) | 5 (6) | 4 (4) | 3 (3) | 4 (4)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 10 (13) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.